CLINICAL TRIAL: NCT07253025
Title: Comparison of Post Operative Pain in Resin-Based and Bio Ceramic Based Root Canal Sealer in Patient Presenting at Peshawar Dental College
Brief Title: Comparison of Post Operative Pain in Resin-Based and Bioceramic Based Root Canal Sealers in Patient Presenting at Peshawar Dental College.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prime Foundation (Other)
Responsible Party: Principal Investigator, Shah Zaman, Docter, Prime Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Prime Foundation Pakistan
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POST OPERATIVE PAIN IN RESIN-BASED ROOT CANAL SEALERS (Other): Patients will be randomly divided into two groups .one group will recived Resin-based sealer (AH Plus)-Group A (90) . Before treatment the patients will be educated that how to complete a visual analog scale (VAS) to evaluate their pain score.
  Interventions: Other: Resin based root canal sealer
- POST OPERATIVE PAIN BIOCERAMIC BASED ROOT CANAL SEALERS (Other): Patients will be randomly divided into two groups. Mineral trioxide aggregate (MTA) fillapex-Group B (90). Before treatment the patients will be educated that how to complete a visual analog scale (VAS) to evaluate their pain score.
  Interventions: Other: Bioceramic based root canal sealer

INTERVENTIONS:
Other: Resin based root canal sealer — Before treatment the patients will be educated that how to complete a visual analog scale (VAS) to evaluate their pain score. Postoperative VAS scores will be recorded after the 24 hours and 48 hours of the treatment for the determination of post-operative pain. All assessment will be recorded on a pre-designed proforma.
  The VAS included a 10 cm straight horizontal line numbered at each centimeter with the following criteria It will be defined on the basis of Visual Analog Score (VAS) after 24 hours in both treatment groups. VAS includes 0-10 numbers, where 0 indicates no pain, and 10 indicates the severe pain. Presence of pain will be validated, if Pain > 3 on VAS.
  Arms: POST OPERATIVE PAIN IN RESIN-BASED ROOT CANAL SEALERS
Other: Bioceramic based root canal sealer — Before treatment the patients will be educated that how to complete a visual analog scale (VAS) to evaluate their pain score. Postoperative VAS scores will be recorded after the 24 hours and 48 hours of the treatment for the determination of post-operative pain. All assessment will be recorded on a pre-designed proforma.
  The VAS included a 10 cm straight horizontal line numbered at each centimeter with the following criteria It will be defined on the basis of Visual Analog Score (VAS) after 24 hours in both treatment groups. VAS includes 0-10 numbers, where 0 indicates no pain, and 10 indicates
  Arms: POST OPERATIVE PAIN BIOCERAMIC BASED ROOT CANAL SEALERS

SUMMARY:
The goal of this clinical trial is to compare the post operative pain in Resin-Based and Bio ceramic based sealers in patients presenting at Peshawar dental college.

Root canal sealer is a material use to avoid gaps between the filling material and root canal Walls, if it is extended beyond canals can cause mild inflammation and post operative pain Hypothesis: There is difference in post operative pain in Resin based and Bio ceramic based sealers in patients presenting at Peshawar dental college.

.Post operative pain:: It will be defined on the basis of Visual Analog Score (VAS) after 24 hours and 48hours in both treatment groups. VAS includes 0-10 numbers, where 0 indicates no pain, and 10 indicates the severe pain. Presence of pain will be validated, if Pain > 3 on VAS.

•The calculated sample size is 180 (90 in each group) Patients will be briefed with information related to the goals, risks, and benefits of the study, and written informed consent form will be taken from all participating patients. To make sure the inclusion criteria are strictly enforced, medical history will be taken. Demographic information like to age, gender, and address will be recorded on a designated proforma. Maxillary or mandibular single-rooted teeth confirmed with symptomatic irreversible pulpitis i.e. normal apical tissues/symptomatic apical periodontitis will be included. Patients will be randomly divided into two groups Resin-based sealer (AH Plus)-Group A (90) and mineral trioxide aggregate (MTA) fillapex-Group B (90) by lottery method. Before treatment the patients will be educated that how to complete a visual analogue scale (VAS) to evaluate their pain score. The VAS included a 10 cm straight horizontal line numbered at each centimetre with the following criteria. Local anaesthetic with 2% lignocaine containing 1:80000 epinephrine will be administered to each patient. A rubber dam will be applied. The endodontic access cavities will be formed with endo access burs. Working length will be established with #10 K file and the root canal will be instrumented with one shape rotary system up to #25.6% under copious irrigation with 3% sodium hypochlorite. Before obturation root canals will be final rinse with 5 ml of 17% EDTA solution. In both treatment groups, the root canal will be dried with paper points and obdurate with cold lateral compaction technique with the help of gutta-percha cones and AH plus /MTA fillapex. Coronal access cavities will be restored with direct composite restorations with the help of dentinal adhesives and universal composite resin. The continuous-wave approach will be used in the AH Plus group, and the single-cone approach will be used in the MTA fillapex. Postoperative VAS scores will be recorded after the 24 hours and 48 hours of the treatment for the determination of post-operative pain. All assessment will be recorded on a pre-designed proforma.

ELIGIBILITY:
Inclusion Criteria:

* Gender Both males and females
* Age Group (18-70) Years
* Patients with Mandibular or Maxillary single-rooted teeth identified with symptomatic irreversible pulpitis either with symptomatic apical periodontitis or normal apical tissues

Exclusion Criteria:

* Patients with immature apices
* Patients with root resorption
* Patients medically compromised, Patients on medications i.e analgesic or anti-inflammatory drugs,
* pregnant/lactating females
* Patient came with flare up pain
* Patients who refused to participate in this study.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Change in the baseline of pain, as measure by the visual analog scale ( VAS) | 24 hours , 48 hours
  Scores are measure on 10 numbers on VAS , where 0 Indicate no pain and 10 Indicate severe pain , presence of pain will be validated, if pain score >3 on VAS scale,

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shah Zaman, BDS, Principal Investigator
Locations (1):
- Peshawar Dental Collge, Peshawar, Khyber Pakhtoon Khawa(KPK)a, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, inform consent, study results
Supporting Information: Study Protocol, ICF
Time Frame: Material will be available 6 months after publication of primary outcomes
Access Criteria: Investigators having studying similar primary outcomes

REFERENCES:
- See also: Parent study Reference — http://www.ijss-sn.com/uploads/2/0/1/5/20153321/09_ijss_sep_21_oa05_-_2021.pdf

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT07253025/Prot_SAP_ICF_000.pdf